CLINICAL TRIAL: NCT06944509
Title: RADIQAL Study (Radiation Dose and Image Quality Trial)
Acronym: RADIQAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IGT-200140-RADIQAL
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: invasive diagnostic procedures; diagnostic coronary angiographies; percutaneous coronary interventions; invasive coronary angiography; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, unblinded, comparative, international, multi-center clinical investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Xres5) (Experimental): treatment with the Azurion system with Xres5
  Interventions: Device: treatment with the Azurion system with Xres5
- Control (ClarityIQ) (Active Comparator): the standard of care (ClarityIQ/Xres4)
  Interventions: Other: Azurion with Clairy IQ

INTERVENTIONS:
Device: treatment with the Azurion system with Xres5 — treatment with the Azurion system with Xres5
  Arms: Intervention (Xres5)
Other: Azurion with Clairy IQ — Azurion system with the standard of care (ClarityIQ/Xres4)
  Arms: Control (ClarityIQ)

SUMMARY:
The Azurion R4.0 is developed by Philips Medical Systems Nederland B.V., a Philips Healthcare company. The Azurion is an interventional X-ray system which is used for live X-ray imaging during invasive cardiac procedures. The proposed Azurion R4.0 includes new x-ray image postprocessing (Xres5) compared to its predecessor, which was equipped with ClarityIQ image post-processing (Xres4).

Azurion R4.0 is a cleared device for EU-MDR regulated countries, submission for FDA510K clearance in the US is pending. Sites in the US will only be activated in the study after FDA clearance.

This is a prospective, randomized, unblinded, comparative, international, multi-center clinical investigation. Randomization will be 1:1 between Xres5 and ClarityIQ (Xres4). Stratification will be performed per site on intended procedure type (based on clinical presentation) and patient BMI.

Primary objective is to demonstrate that in coronary procedures, Xres5 can reduce overall patient radiation dose compared to the current ClarityIQ without affecting procedural performance.

It is expected that 824 subjects are necessary to collect sufficient data for the evaluation of the objectives of this clinical study. The enrollment period is expected to last for 12 months. The study will be executed in Spain, Czech republic, Denmark and the US.

DETAILED DESCRIPTION:
The study procedures consist of three main steps: 1) patient screening and written informed consent, 2) baseline assessment and randomization and 3) treatment with the Azurion system with Xres5 [intervention] or the standard of care (ClarityIQ/Xres4) [control]. Patients will be randomly assigned to either the intervention group or the control group (using the standard of care) in a 1:1 ratio. The coronary procedure will be conducted as per institutional standards and at the discretion of the operator, but the standard image processing will be based on the randomization result. If randomized to the intervention group (Xres5), it will always be possible for the operator to cross over to the standard of care imaging processing (Clarity IQ). For the study sites in EU the primary staff in the intervention room will be wearing electronic staff dosimeters which will log the radiation exposure per staff member per procedure.

After the procedure, characteristics of the patient and procedure are captured in an eCRF. The imaging runs will be uploaded in the cloud after de-identification. After the study the radiation dose (DAP and Air Kerma) will be read out from the system.

The study procedures will end after the coronary procedure is completed. There will be no modifications in the standard of care patient treatment or follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be undergoing a diagnostic angiography and/or coronary intervention /elective PCI.
* Subject is able to give written informed consent.
* Subject is 18 years of age or older, or of legal age to give informed consent per state or national law.

Exclusion Criteria:

* Subject with known contrast allergy that cannot be adequately premedicated.
* Subject with previous contraindication for diagnostic angiography and/or diagnostic/elective PCI.
* Subject participates in a potentially confounding drug or device study during the course of the study.
* All vulnerable subjects such as pregnant or breast-feeding women, or any other subject who meets an exclusion criteria according to applicable national laws, if any.
* Subject unwilling or unable to comply with the protocol and/or unable to understand verbal and/or written informed consent.
* Expected use of non-standard contrast concentrations (e.g. dilution of contrast).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient radiation dose and procedural performance (ClarityIQ vs Xres5) | during study procedure
  - Cumulative Dose Area Product (DAP) [Gycm2]
  Total patient group - All procedure types
Patient radiation dose and procedural performance (ClarityIQ vs Xres5) | during study procedure
  - Cumulative Air Kerma (AK) [Gy]
  Total patient group - All procedure types
Patient radiation dose and procedural performance (ClarityIQ vs Xres5) | during study procedure
  - Time System in Use* [minutes]
  Total patient group - All procedure types

SECONDARY OUTCOMES:
Patient radiation dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Cumulative DAP [Gycm2]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedures types
Patient radiation dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Air Kerma [Gy]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedures types
Patient radiation dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Time System in Use* [minutes]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedures types
Patient radiation dose and procedural performance in diagnostic procedures (ClarityIQ vs Xres5) | During study procedure
  - Cumulative DAP [Gycm2]
  Total patient group - ICA procedures
Patient radiation dose and procedural performance in diagnostic procedures (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Air Kerma [Gy]
  Total patient group - ICA procedures
Patient radiation dose and procedural performance in diagnostic procedures (ClarityIQ vs Xres5) | During study procedure
  - Time System in Use* [minutes]
  Total patient group - ICA procedures
Patient radiation dose and procedural performance in interventional procedures (ClarityIQ vs Xres5) | During study procedure
  - Cumulative DAP [Gycm2]
  Total patient group - PCI and ICA+PCI procedures
Patient radiation dose and procedural performance in interventional procedures (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Air Kerma [Gy]
  Total patient group - PCI and ICA+PCI procedures
Patient radiation dose and procedural performance in interventional procedures (ClarityIQ vs Xres5) | During study procedure
  - Time System in Use* [minutes]
  Total patient group - PCI and ICA+PCI procedures
Coronary Cine Radiation Dose and procedural performance (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Cine Air Kerma [Gy]
  Total patient group - All procedure types - Coronary Cine Data
Coronary Cine Radiation Dose and procedural performance (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Cine DAP [Gycm2]
  Total patient group - All procedure types - Coronary Cine Data
Coronary Cine Radiation Dose and procedural performance (ClarityIQ vs Xres5) | During study procedure
  - Time System in Use* [minutes]
  Total patient group - All procedure types - Coronary Cine Data
Coronary Cine Radiation Dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Cine Air Kerma [Gy]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedure types - Coronary Cine Data
Coronary Cine Radiation Dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Cumulative Cine DAP [Gycm2]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedure types - Coronary Cine Data
Coronary Cine Radiation Dose and procedural performance - High BMI (ClarityIQ vs Xres5) | During study procedure
  - Time System in Use* [minutes]
  High BMI patients (BMI ≥ 30 kg/m2) - All procedure types - Coronary Cine Data
Ultra-low dose cine fluoro rate (Xres5) | During study procedure
  - Air Kerma rate per acquisitions [mGy/minutes]
  Xres5 cases - Total Patient group - All procedure types

OTHER OUTCOMES:
Staff radiation dose (ClarityIQ vs Xres5) | During study procedure
  - Deep dose Hp(10) [mSv]
  Total Patient group - All procedure types
Staff radiation dose (ClarityIQ vs Xres5) | During study procedure
  - Skin dose Hp(0.07) [mSv]
  Total Patient group - All procedure types
Iodine contrast volume administered (ClarityIQ vs Xres5) | During study procedure
  - Iodinated contrast volume [ml]
  Total Patient group - All procedure types
Patient Radiation Dose - Projection Angles (ClarityIQ vs Xres5) | During study procedure
  - DAP per run [Gycm2]
  Total Patient group - All procedure types
Patient Radiation Dose - Projection Angles (ClarityIQ vs Xres5) | During study procedure
  - Air Kerma per run [Gy]
  Total Patient group - All procedure types

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - NYP Columbia, New York, New York
- University Hospital Královské Vinohrady, Prague, Czechia
- Aarhus university hospital, Aarhus, Denmark
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philips Medical Systems Nederland B.V., "Safety and feasibility study with a new X-ray processing algorithm (Xres5) for coronary procedures"
- [Background] Gislason-Lee AJ, Keeble C, Malkin CJ, Egleston D, Bexon J, Kengyelics SM, Blackman D, Davies AG. Impact of latest generation cardiac interventional X-ray equipment on patient image quality and radiation dose for trans-catheter aortic valve implantations. Br J Radiol. 2016 Nov;89(1067):20160269. doi: 10.1259/bjr.20160269. Epub 2016 Sep 29. PMID 27610932
- [Background] Nakamura S, Kobayashi T, Funatsu A, Okada T, Mauti M, Waizumi Y, Yamada S. Patient radiation dose reduction using an X-ray imaging noise reduction technology for cardiac angiography and intervention. Heart Vessels. 2016 May;31(5):655-63. doi: 10.1007/s00380-015-0667-z. Epub 2015 Apr 4. PMID 25840815
- [Background] Hruby A, Hu FB. The Epidemiology of Obesity: A Big Picture. Pharmacoeconomics. 2015 Jul;33(7):673-89. doi: 10.1007/s40273-014-0243-x. PMID 25471927
- [Background] Smith IR, Rivers JT. Measures of radiation exposure in cardiac imaging and the impact of case complexity. Heart Lung Circ. 2008 Jun;17(3):224-31. doi: 10.1016/j.hlc.2007.10.004. Epub 2008 Jan 31. PMID 18242136
- [Background] Cusma JT, Bell MR, Wondrow MA, Taubel JP, Holmes DR Jr. Real-time measurement of radiation exposure to patients during diagnostic coronary angiography and percutaneous interventional procedures. J Am Coll Cardiol. 1999 Feb;33(2):427-35. doi: 10.1016/s0735-1097(98)00591-9. PMID 9973023
- [Background] Fetterly KA, Lennon RJ, Bell MR, Holmes DR Jr, Rihal CS. Clinical determinants of radiation dose in percutaneous coronary interventional procedures: influence of patient size, procedure complexity, and performing physician. JACC Cardiovasc Interv. 2011 Mar;4(3):336-43. doi: 10.1016/j.jcin.2010.10.014. PMID 21435613